CLINICAL TRIAL: NCT02394561
Title: A 24-week, Multicenter, proSpective stUdy to Evaluate the PASI 90 Clinical Response Rate and the Safety PRofile of sEcukinuMab 300 mg in Cw6-negativE and Cw6-positive Patients With Moderate to Severe Chronic Plaque-type Psoriasis (SUPREME)
Acronym: SUPREME
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAIN457AIT01
Record Dates: First submitted 2015-02-25; First posted 2015-03-20 (Estimated); Results first posted 2019-04-23 (Actual); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Plaque Type Psorisis
MeSH Terms: interventions — secukinumab

STUDY DESIGN:
Intervention Model Description: Arms represent stratification of Cw6 positive and Cw6 negative patients
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cw6-positive AIN457 300 mg (Experimental): Stratified to Cw6 positive cohort. Investigators and patients were blinded to Cw6 results. All patients were treated according to an induction regimen of two injections of secukinumab 150 mg a week for five weeks starting at baseline (week 0), followed by a maintenance period of two injections per month. At week 16, patients achieving PASI 50 response were eligible to continue on secukinumab for an additional 8 weeks in CORE. Eligible patients with at least a PASI 75 response were included in the extension phase, up to 72 weeks
  Interventions: Biological: Secukinumab
- Cw6-negative AIN457 300 mg (Experimental): Stratified to Cw6 negative cohort. Investigators and patients were blinded to Cw6 results. All patients were treated according to an induction regimen of two injections of secukinumab 150 mg a week for five weeks starting at baseline (week 0), followed by a maintenance period of two injections per month. At week 16, patients achieving PASI 50 response were eligible to continue on secukinumab for an additional 8 weeks in CORE. Eligible patients with at least a PASI 75 response were included in the extension phase, up to 72 weeks
  Interventions: Biological: Secukinumab

INTERVENTIONS:
Biological: Secukinumab — Secukinumab was supplied as 150 mg solution in pre-filled syringe for subcutaneous injection
  Other Names: AIN457

SUMMARY:
A study to evaluate the differences in the efficacy and safety of secukinumab between Cw6-negative and Cw6-positive patients with moderate to severe plaque-type psoriasis

DETAILED DESCRIPTION:
Biological agents represent the most advanced type of treatment for psoriasis. Secukinumab is a human monoclonal anti IL-17A antibody that binds to human IL-17A and neutralizes its bioactivity by inhibiting IL17A produced by both Th17 cells and those of the innate immune system, thus providing complete anti IL17A blockage. Targeting IL-17A has the potential to reduce autoimmune inflammation while leaving other immune functions undisturbed. While targeting of Th1-promoting or Th17-promoting cytokines affects critical mediators such as IFN-γ, IL-22 and IL-21, selective targeting of IL-17A leaves these Th1/17 activities, as well as certain protective functions of innate cells intact. Furthermore, as a fully human monoclonal antibody, secukinumab should reduce immunogenic risks compared to current or emerging antibody therapies that are not fully human.

Many recent studies have shown that highly selective biologic drugs are not effective in every patient and that variations in the genome can be associated with different clinical responses or side effects to a given drug. The PSORS1 locus on chromosome 6p is generally understood to confer the most risk for psoriasis. A specific allele for this locus, HLA C*06, is present in about 60% of psoriatic patient cases. Data linking secukinumab efficacy to a particular genetic marker are lacking.

Recent research has revealed a marked difference in the proportion of PASI 90 achievers at 12 weeks between Cw6-positive and Cw6-negative patients (85.7% vs 56.5%) treated with ustekinumab (Talamonti M et al. 2013) and a greater efficacy of anti-TNFα drugs in CW6 negative patients (Galli et al. 2013).Unlike anti-IL-12/23 agents, secukinumab inhibits IL-17 produced by both Th17 cells after presentation by antigen presenting cells (in this case Cw6) and cells of the innate immune system whose activation does not require antigen presentation. Providing a drug that is equally effective on both Cw6-negative and Cw6-positive patients would be an important clinical accomplishment and would eliminate the need for costly HLA-Cw6 tests. The choice of a cohort study would therefore seem appropriate for this clinical context.

The purpose of this study was to explore the different efficacy and safety profile of secukinumab 300 mg in patients with moderate to severe chronic plaque-type psoriasis, stratified for the presence of HLA-C*06, whose determination was blinded for patients and investigators. The study was conducted both on anti-TNFα-naïve and anti-TNFα failure patients and also stratified for TNFα - 308 polymorphism, BMI, smoking and metabolic syndrome, among others.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must have been able to understand and communicate with the investigator and to comply with the requirements of the study and must have given a written, signed and dated informed consent before any study related activity was performed.
2. Men or women at least 18 years of age at time of screening.
3. Diagnosis of moderate to severe chronic plaque-type psoriasis for at least 6 months (including concomitant psoriatic arthritis as per the Classification Criteria for Psoriatic Arthritis criteria [CASPAR]).
4. Moderate to severe psoriasis as defined at enrollment by:

   * PASI score ≥ 10 or
   * PASI score > 5 but < 10 and DLQI ≥10
5. Patients that are candidates for systemic therapy, whether treatment naïve or after failed response to other systemic therapy (i.e. cyclosporine, methotrexate and PUVA) or to an anti-TNFα (or is intolerant and/or has a contraindication to these).

Exclusion criteria

1. Forms of psoriasis other than chronic plaque-type (e.g., pustular, erythrodermic and guttate psoriasis).
2. Cyclosporine or methotrexate therapy within 4 weeks prior to Day 1.
3. Anti-TNFα therapy within timelines depending on drug half-life.
4. Previous exposure to secukinumab or any other biologic drug directly targeting IL-17 or the IL-17 receptor.
5. Previous exposure to ustekinumab or any other biologic drug for the treatment of psoriasis that was not anti-TNFα therapy.
6. Intravenous or intramuscular steroids within 2 weeks prior to screening and during screening.
7. Ongoing use of corticosteroid topical treatments or UV therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 434 (Actual)
Dates: Start 2015-04-10 (Actual); Primary Completion 2017-06-08 (Actual); Study Completion 2017-06-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (40):
- Italy (40):
  - Novartis Investigative Site, Milan, (MI)
  - Novartis Investigative Site, Ancona, AN
  - Novartis Investigative Site, L’Aquila, AQ
  - Novartis Investigative Site, Bari, BA
  - Novartis Investigative Site, Bergamo, BG
  - Novartis Investigative Site, Benevento, BN
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Brindisi, BR
  - Novartis Investigative Site, Brescia, BS
  - Novartis Investigative Site, Cagliari, CA
  - Novartis Investigative Site, Chieti, CH
  - Novartis Investigative Site, Catania, CT
  - Novartis Investigative Site, Catanzaro, CZ
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Grosseto, GR
  - Novartis Investigative Site, Lecce, LE
  - Novartis Investigative Site, Terracina, LT
  - Novartis Investigative Site, Lucca, LU
  - Novartis Investigative Site, Macerata, MC
  - Novartis Investigative Site, Messina, ME
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, San Donato Milanese, MI
  - Novartis Investigative Site, Mantova, MN
  - Novartis Investigative Site, Modena, MO
  - Novartis Investigative Site, Padua, PD
  - Novartis Investigative Site, Perugia, PG
  - Novartis Investigative Site, Pisa, PI
  - Novartis Investigative Site, Parma, PR
  - Novartis Investigative Site, Pavia, PV
  - Novartis Investigative Site, Reggio Emilia, RE
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Siena, SI
  - Novartis Investigative Site, Torino, TO
  - Novartis Investigative Site, Erice, TP
  - Novartis Investigative Site, Terni, TR
  - Novartis Investigative Site, Trieste, TS
  - Novartis Investigative Site, Udine, UD
  - Novartis Investigative Site, Verona, VR
  - Novartis Investigative Site, Napoli

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Five hundred thirty participants were screened and 434 entered the CORE Phase. However, there were 3 patients without Cw6 assessment which was necessary for stratification to the two arms, therefore 431 were considered enrolled.
Period: CORE Phase
Arm/Group | Cw6-positive AIN457 300 mg | Cw6-negative AIN457 300 mg
Started | 185 | 246
Full Analysis Set | 185 | 246
Safety Set | 185 | 246
ITT Set | 184 | 246
Completed | 172 | 227
Not Completed | 13 | 19
Not completed — Adverse Event | 7 | 9
Not completed — Death | 0 | 1
Not completed — Pregnancy | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Physician Decision | 1 | 1
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Lack of Efficacy | 1 | 6
Period: Extension Phase
Arm/Group | Cw6-positive AIN457 300 mg | Cw6-negative AIN457 300 mg
Started | 162 | 219
Completed | 151 | 207
Not Completed | 11 | 12
Not completed — Adverse Event | 6 | 1
Not completed — Death | 0 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Physician Decision | 0 | 2
Not completed — Withdrawal by Subject | 0 | 5
Not completed — Lack of Efficacy | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cw6-positive AIN457 300 mg | Cw6-negative AIN457 300 mg | Total
Number analyzed (Participants) | 185 | 246 | 431
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.71 (13.148) | 47.18 (12.919) | 45.26 (13.189)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 62 | 122
  Male | 125 | 184 | 309
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 184 | 241 | 425
  Asian | 0 | 1 | 1
  Native American | 0 | 1 | 1
  Unknown | 0 | 2 | 2
  Other | 1 | 1 | 2
Time since first diagnosis of psoriasis [Mean (Standard Deviation); unit: years] | 19.63 (12.489) | 17.46 (11.343) | 18.39 (11.883)

OUTCOME MEASURES:

1. Primary Outcome: Percentage (%) of Patients Who Reach Psoriasis Area Severity Index (PASI) 90 at 16 Weeks - LOCF Approach (ITT Set)
Description: PASI (Langley et al 2015) combines the assessment of the severity of lesions and the area affected into a single score with a range of 0 (no disease) to 72 (maximal disease). The PASI was assessed at all visits in CORE and extension phases. PASI 90 response: patients achieving ≥ 90% improvement (reduction) in PASI score compared to baseline are defined as PASI 90 responders.
Time Frame: Baseline up to 16 weeks
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cw6-positive AIN457 300 mg | Cw6-negative AIN457 300 mg
Number analyzed (Participants) | 184 | 246
percentage of participants | 80.4 [74.0 to 85.9] | 81.7 [76.3 to 86.3]
Statistical Analysis 1: Comparison: Cw6-negative AIN457 300 mg; Test type: Non-Inferiority — The difference in percentage of patients achieving PASI 90 response between the Cw6-positive cohort and the Cw6-negative cohort was H0 = Cw6-positive minus Cw6-negative ≥0.12 and HA = Cw6-positive minus Cw6-negative was < 0.12. The percentage of PASI 90 response by cohort as well as the difference between cohort together with 97.5% upper CI was provided using Clopper Pearson CI method; difference = -1.3, 95% CI 2-sided [-8.8 to 6.2]

2. Secondary Outcome: Percentage (%) of Patients With IGA 0/1, PASI 50, PASI 75, PASI 90, PASI 100 Responders by Visit - LOCF Approach (ITT Set)
Description: IGA mod 2011 scale measures severity of the psoriasis on a five-point scale ranging from 0 (no disease, 'clear') to 4 ('very severe'). PASI 50,75,90,100 represent: patients achieving ≥ 50% improvement (reduction) in PASI score compared to baseline, ≥ 75% improvement (reduction), ≥ 90% improvement (reduction) and PASI 100 response/remission: complete clearing of psoriasis (PASI=0).
Time Frame: Baseline up to approximately 72 weeks
Population: Number of patients varied across visits
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Difference in % (Cw6-pos vs Cw6-neg): Difference in percentages of the two cohorts in IGA 0/1 and PASI 50, 75, 90,100 at all time points.
Arm/Group | Cw6-positive AIN457 300 mg | Cw6-negative AIN457 300 mg | Difference in % (Cw6-pos vs Cw6-neg)
Number analyzed (Participants) | 184 | 246 | 430
percentage of participants
  W1 IGA 0/1: number analyzed (Participants) | 178 | 240 | 418
  W1 IGA 0/1 | 2.2 [0.62 to 5.65] | 2.1 [0.68 to 4.79] | 0.16 [-2.86 to 3.75]
  W1 PASI 50: number analyzed (Participants) | 179 | 240 | 419
  W1 PASI 50 | 13.4 [8.78 to 19.29] | 12.1 [8.24 to 16.89] | 1.32 [-5.02 to 8.09]
  W1 PASI 75: number analyzed (Participants) | 179 | 240 | 419
  W1 PASI 75 | 2.2 [0.61 to 5.62] | 0.4 [0.01 to 2.30] | 1.82 [-0.52 to 5.20]
  W2 IGA 0/1 | 8.7 [5.05 to 13.74] | 6.9 [4.08 to 10.83] | 1.79 [-3.29 to 7.36]
  W2 PASI 50: number analyzed (Participants) | 184 | 245 | 430
  W2 PASI 50 | 44.0 [36.73 to 51.51] | 44.5 [38.16 to 50.95] | -0.47 [-9.84 to 8.98]
  W2 PASI 75: number analyzed (Participants) | 184 | 245 | 430
  W2 PASI 75 | 15.8 [10.82 to 21.84] | 10.2 [6.71 to 14.69] | 5.56 [-0.80 to 12.32]
  W2 PASI 90: number analyzed (Participants) | 184 | 245 | 430
  W2 PASI 90 | 3.3 [1.21 to 6.96] | 2.4 [0.90 to 5.25] | 0.81 [-2.49 to 4.71]
  W2 PASI 100: number analyzed (Participants) | 184 | 245 | 430
  W2 PASI 100 | 0.5 [0.01 to 2.99] | 0.4 [0.01 to 2.25] | 0.14 [-1.78 to 2.63]
  W3 IGA 0/1 | 24.5 [18.43 to 31.32] | 21.1 [16.21 to 26.78] | 3.32 [-4.58 to 11.46]
  W3 PASI 50: number analyzed (Participants) | 184 | 245 | 429
  W3 PASI 50 | 76.1 [69.26 to 82.06] | 71.8 [65.76 to 77.38] | 4.25 [-4.23 to 12.40]
  W3 PASI 75: number analyzed (Participants) | 184 | 245 | 429
  W3 PASI 75 | 38.6 [31.52 to 46.03] | 34.3 [28.36 to 40.60] | 4.30 [-4.81 to 13.46]
  W3 PASI 90: number analyzed (Participants) | 184 | 245 | 429
  W3 PASI 90 | 13.0 [8.54 to 18.78] | 11.4 [7.73 to 16.09] | 1.61 [-4.55 to 8.19]
  W3 PASI 100: number analyzed (Participants) | 184 | 245 | 429
  W3 PASI 100 | 2.7 [0.89 to 6.23] | 2.4 [0.90 to 5.25] | 0.27 [-2.92 to 4.00]
  W4 IGA 0/1 | 42.4 [35.15 to 49.88] | 39.8 [33.67 to 46.25] | 2.55 [-6.75 to 11.89]
  W4 PASI 50 | 87.5 [81.84 to 91.91] | 87.4 [82.59 to 91.27] | 0.10 [-6.51 to 6.31]
  W4 PASI 75 | 61.4 [53.97 to 68.48] | 57.3 [50.88 to 63.58] | 4.10 [-5.29 to 13.28]
  W4 PASI 90 | 27.7 [21.39 to 34.78] | 22.0 [16.94 to 27.65] | 5.77 [-2.40 to 14.10]
  W4 PASI 100 | 10.3 [6.33 to 15.66] | 9.8 [6.35 to 14.17] | 0.57 [-5.09 to 6.66]
  W8 IGA 0/1 | 72.3 [65.22 to 78.61] | 73.2 [67.17 to 78.60] | -0.89 [-9.48 to 7.47]
  W8 PASI 50 | 95.7 [91.61 to 98.10] | 95.1 [91.63 to 97.45] | 0.53 [-3.97 to 4.59]
  W8 PASI 75 | 84.8 [78.76 to 89.64] | 85.0 [79.87 to 89.18] | -0.18 [-7.26 to 6.53]
  W8 PASI 90 | 61.4 [53.97 to 68.48] | 60.6 [54.16 to 66.72] | 0.84 [-8.46 to 10.01]
  W8 PASI 100 | 34.8 [27.93 to 42.14] | 34.6 [28.63 to 40.86] | 0.23 [-8.72 to 9.34]
  WK12 IGA 0/1 | 81.0 [74.55 to 86.38] | 81.7 [76.30 to 86.33] | -0.73 [-8.36 to 6.57]
  WK12 PASI 50 | 97.3 [93.77 to 99.11] | 97.2 [94.23 to 98.85] | 0.13 [-3.65 to 3.43]
  WK12 PASI 75 | 92.9 [88.22 to 96.18] | 90.7 [86.30 to 93.98] | 2.28 [-3.27 to 7.46]
  WK12 PASI 90 | 72.8 [65.79 to 79.11] | 73.6 [67.60 to 78.98] | -0.75 [-9.30 to 7.56]
  WK12 PASI 100 | 49.5 [42.02 to 56.91] | 43.9 [37.60 to 50.35] | 5.55 [-3.93 to 14.94]
  WK16 IGA 0/1 | 85.3 [79.37 to 90.10] | 86.2 [81.23 to 90.23] | -0.85 [-7.79 to 5.70]
  WK16 PASI 50 | 97.8 [94.53 to 99.40] | 98.8 [96.48 to 99.75] | -0.95 [-4.33 to 1.70]
  WK16 PASI 75 | 94.0 [89.56 to 96.98] | 93.1 [89.17 to 95.92] | 0.93 [-4.16 to 5.60]
  WK16 PASI 90 | 80.4 [73.96 to 85.90] | 81.7 [76.30 to 86.33] | -1.27 [-8.94 to 6.08]
  WK16 PASI 100 | 59.2 [51.77 to 66.41] | 53.3 [46.81 to 59.62] | 5.99 [-3.49 to 15.24]
  WK20 IGA0/1 | 87.0 [81.22 to 91.46] | 87.4 [82.59 to 91.27] | -0.44 [-7.11 to 5.83]
  WK20 PASI 50 | 97.8 [94.53 to 99.40] | 97.6 [94.77 to 99.10] | 0.27 [-3.27 to 3.34]
  WK20 PASI 75 | 94.6 [90.23 to 97.36] | 92.7 [88.68 to 95.61] | 1.88 [-3.14 to 6.53]
  WK20 PASI 90 | 81.0 [74.55 to 86.38] | 81.7 [76.30 to 86.33] | -0.73 [-8.36 to 6.57]
  WK20 PASI 100 | 59.8 [52.32 to 66.93] | 57.3 [50.88 to 63.58] | 2.47 [-6.93 to 11.71]
  WK24 IGA 0/1 | 89.7 [84.34 to 93.67] | 85.4 [80.32 to 89.54] | 4.31 [-2.21 to 10.45]
  WK24 PASI 50 | 97.3 [93.77 to 99.11] | 97.2 [94.23 to 98.85] | 0.13 [-3.65 to 3.43]
  WK24 PASI 75 | 94.6 [90.23 to 97.36] | 93.1 [89.17 to 95.92] | 1.48 [-3.51 to 6.07]
  WK24 PASI 90 | 84.2 [78.16 to 89.18] | 83.3 [78.08 to 87.77] | 0.91 [-6.35 to 7.79]
  WK24 PASI 100 | 62.0 [54.52 to 69.00] | 61.4 [54.99 to 67.50] | 0.57 [-8.71 to 9.71]
  WK36 IGA 0/1: number analyzed (Participants) | 161 | 219 | 380
  WK36 IGA 0/1 | 91.9 [86.59 to 95.63] | 90.9 [86.25 to 94.33] | 1.06 [-5.06 to 6.68]
  WK36 PASI 50: number analyzed (Participants) | 161 | 219 | 380
  WK36 PASI 50 | 98.8 [95.58 to 99.85] | 99.1 [96.74 to 99.89] | -0.33 [-3.57 to 2.19]
  WK36 PASI 75: number analyzed (Participants) | 161 | 219 | 380
  WK36 PASI 75 | 94.4 [89.65 to 97.41] | 95.0 [91.19 to 97.47] | -0.57 [-5.75 to 4.00]
  WK36 PASI 90: number analyzed (Participants) | 161 | 219 | 380
  WK36 PASI 90 | 88.8 [82.91 to 93.24] | 84.0 [78.48 to 88.61] | 4.80 [-2.39 to 11.54]
  WK36 PASI 100: number analyzed (Participants) | 161 | 219 | 380
  WK36 PASI 100 | 65.8 [57.96 to 73.12] | 64.4 [57.65 to 70.72] | 1.45 [-8.27 to 10.95]
  WK48 IGA 0/1: number analyzed (Participants) | 115 | 159 | 274
  WK48 IGA 0/1 | 87.8 [80.42 to 93.18] | 86.8 [80.52 to 91.63] | 1.03 [-7.43 to 8.82]
  WK48 PASI 50: number analyzed (Participants) | 115 | 159 | 274
  WK48 PASI 50 | 98.3 [93.86 to 99.79] | 98.1 [94.59 to 99.61] | 0.15 [-4.41 to 3.88]
  WK48 PASI 75: number analyzed (Participants) | 115 | 159 | 274
  WK48 PASI 75 | 93.9 [87.86 to 97.52] | 91.2 [85.67 to 95.10] | 2.72 [-4.18 to 8.98]
  WK48 PASI 90: number analyzed (Participants) | 115 | 159 | 274
  WK48 PASI 90 | 84.3 [76.40 to 90.45] | 80.5 [73.48 to 86.35] | 3.84 [-5.59 to 12.64]
  WK48 PASI 100: number analyzed (Participants) | 115 | 159 | 274
  WK48 PASI 100 | 68.7 [59.38 to 77.02] | 61.6 [53.60 to 69.23] | 7.06 [-4.44 to 18.02]
  WK60 IGA 0/1: number analyzed (Participants) | 80 | 118 | 198
  WK60 IGA 0/1 | 87.5 [78.21 to 93.84] | 83.9 [76.00 to 90.02] | 3.60 [-6.97 to 13.09]
  WK60 PASI 50: number analyzed (Participants) | 80 | 119 | 199
  WK60 PASI 50 | 96.3 [89.43 to 99.22] | 95.0 [89.35 to 98.13] | 1.29 [-5.94 to 7.34]
  WK60 PASI 75: number analyzed (Participants) | 80 | 119 | 199
  WK60 PASI 75 | 90.0 [81.24 to 95.58] | 89.9 [83.05 to 94.68] | 0.08 [-9.42 to 8.37]
  WK60 PASI 90: number analyzed (Participants) | 80 | 119 | 199
  WK60 PASI 90 | 82.5 [72.38 to 90.09] | 74.8 [66.01 to 82.30] | 7.71 [-4.27 to 18.58]
  WK60 PASI 100: number analyzed (Participants) | 80 | 119 | 199
  WK60 PASI 100 | 65.0 [53.52 to 75.33] | 56.3 [46.91 to 65.37] | 8.70 [-5.19 to 21.80]
  WK72 IGA 0/1: number analyzed (Participants) | 41 | 60 | 101
  WK72 IGA 0/1 | 85.4 [70.83 to 94.43] | 80.0 [67.67 to 89.22] | 5.37 [-10.7 to 19.47]
  WK72 PASI 50: number analyzed (Participants) | 41 | 61 | 102
  WK72 PASI 50 | 92.7 [80.08 to 98.46] | 93.4 [84.05 to 98.18] | -0.76 [-13.5 to 9.55]
  WK72 PASI 75: number analyzed (Participants) | 41 | 61 | 102
  WK72 PASI 75 | 85.4 [70.83 to 94.43] | 88.5 [77.78 to 95.26] | -3.16 [-18.1 to 9.79]
  WK72 PASI 90: number analyzed (Participants) | 41 | 61 | 102
  WK72 PASI 90 | 75.6 [59.70 to 87.64] | 73.8 [60.93 to 84.20] | 1.84 [-15.8 to 17.98]
  WK72 PASI 100: number analyzed (Participants) | 41 | 61 | 102
  WK72 PASI 100 | 58.5 [42.11 to 73.68] | 50.8 [37.70 to 63.86] | 7.72 [-11.7 to 26.08]

3. Secondary Outcome: Percent Mean Changes From Baseline in IGA Mod 2011 Between Cohorts at Each Time Point (LOCF) (ITT)
Description: IGA mod 2011 scale measures severity of the psoriasis on a five-point scale ranging from 0 (no disease, 'clear') to 4 ('very severe').
Time Frame: Baseline up to approximately 72 weeks
Population: The number of patients across visits varied
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Cw6-positive AIN457 300 mg | Cw6-negative AIN457 300 mg
Number analyzed (Participants) | 184 | 246
percent change
  W1: number analyzed (Participants) | 178 | 240
  W1 | -8.5 (16.08) | -7.3 (17.04)
  W2 | -22.4 (22.73) | -21.6 (22.72)
  W3 | -38.0 (25.45) | -36.5 (27.20)
  W4 | -49.6 (29.36) | -49.5 (29.24)
  W8 | -71.2 (28.60) | -71.2 (28.91)
  W12 | -78.7 (27.31) | -79.0 (25.37)
  W16 | -84.1 (24.52) | -83.3 (22.97)
  W20 | -85.3 (24.26) | -84.5 (23.80)
  W24 | -86.2 (25.17) | -84.1 (26.34)
  W36: number analyzed (Participants) | 161 | 219
  W36 | -88.6 (22.34) | -87.6 (23.82)
  W48: number analyzed (Participants) | 115 | 159
  W48 | -86.2 (25.75) | -84.9 (26.06)
  W60: number analyzed (Participants) | 80 | 118
  W60 | -83.3 (28.44) | -81.0 (26.97)
  W72: number analyzed (Participants) | 41 | 60
  W72 | -79.1 (32.92) | -75.8 (29.58)

4. Secondary Outcome: Median Time to Reach PASI 90 and 75 (ITT)
Description: Time in days to reach PASI scores of 90 and 75.
Time Frame: Baseline up to approximately 72 weeks
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Cw6-positive AIN457 300 mg | Cw6-negative AIN457 300 mg
Number analyzed (Participants) | 184 | 246
days
  PASI 90 | 57 [30 to 89] | 58 [55 to 92]
  PASI 75 | 29 [22 to 57] | 29 [22 to 57]
Statistical Analysis 1: Comparison: Cw6-positive AIN457 300 mg vs Cw6-negative AIN457 300 mg; Test type: Other — difference between cohorts for PASI 90 using Kaplan-Meier estimate; p = 0.1295, Log Rank
Statistical Analysis 2: Comparison: Cw6-positive AIN457 300 mg vs Cw6-negative AIN457 300 mg; Test type: Other; p = 0.4470, Log Rank — difference between cohorts for PASI 75 using Kaplan-Meier estimate

5. Secondary Outcome: Change From Baseline in the Dermatology Life Quality Index (DLQI) (LOCF) (FAS)
Description: The DLQI total score was calculated by summing the score of each domain resulting in a maximum of 30 and a minimum of 0. The higher the score, the more Quality of Life was impaired. Meaning of DLQI Scores: 0-1 = no effect at all on patient's life, 2-5 = small effect on patient's life, 6-10 = moderate effect on patient's life, 11-20= very large effect on patient's life, 21-30 = extremely large effect on patient's life. It was pre-specified that results would be presented for all patients, not by cohort
Time Frame: Baseline up to approximatly 72 weeks
Population: Number of patients varied across visits. Both arms were combined because there is no clinical rationale to show a difference between the cohorts. Cw6 status does not have any impact on Quality of Life.
Measure: Mean (Standard Deviation); unit: numbers in a score
Groups:
- All Patients: All patients in the Safety Set.
Arm/Group | All Patients
Number analyzed (Participants) | 431
numbers in a score
  Week 16: number analyzed (Participants) | 386
  Week 16 | -8.5 (6.79)
  Week 24: number analyzed (Participants) | 420
  Week 24 | -8.8 (7.05)
  Week 48: number analyzed (Participants) | 384
  Week 48 | -8.9 (7.13)
  Week 72: number analyzed (Participants) | 215
  Week 72 | -8.3 (6.70)
Statistical Analysis 1: Comparison: All Patients; Test type: Superiority; p < .0001, Wilcoxon (Mann-Whitney); At all time points

6. Secondary Outcome: Change From Baseline in Mean Scores of HAD-A and HAD-D (Anxiety and Depression) (LOCF) (FAS)
Description: The Hospital Anxiety and Depression Scale (HADS) is a fourteen-item scale.. Seven of the items relate to anxiety and seven relate to depression. This outcome measure was specifically developed to avoid reliance on aspects of these conditions that are also common somatic symptoms of illness, for example fatigue and insomnia or hypersomnia. Calculations of scores: each of the 14 items was rated on a 4-point scale. All items except 7 and 10 were scored as Yes, definitely = 3, Yes, sometimes = 2, No, not much = 1, to No, not at all = 0. Items 7 and 10 were scored as Yes, definitely = 0 to No, not at all = 3 in the reverse order. The HADS consisted of two sub-scores: the HAD-A (anxiety) and HAD-D (depression); each sub-score ranged from 0 to 21 points; scores ≥11 = presence of anxious or depressive disorders; scores between 8-10 points = borderline abnormal, and scores of ≤7 = disorder was not present. It was pre-specified that results would be presented for all patients, not by cohort
Time Frame: Baseline up approximately 72 weeks
Population: Number of patients varies by visit. Both arms were combined because there is no clinical rationale to show a difference between the cohorts. Cw6 status does not have any impact on anxiety and depression.
Measure: Mean (Standard Deviation); unit: numbers on a scale
Arm/Group | All Patients
Number analyzed (Participants) | 431
numbers on a scale
  W16 Anxiety: number analyzed (Participants) | 388
  W16 Anxiety | -1.7 (3.37)
  W24 Anxiety: number analyzed (Participants) | 420
  W24 Anxiety | -2.0 (3.38)
  W48 Anxiety: number analyzed (Participants) | 384
  W48 Anxiety | -2.5 (3.67)
  W72 Anxiety: number analyzed (Participants) | 214
  W72 Anxiety | -2.3 (3.44)
  W16 Depression: number analyzed (Participants) | 388
  W16 Depression | -1.3 (3.19)
  W24 Depression: number analyzed (Participants) | 420
  W24 Depression | -1.4 (3.22)
  W48 Depression: number analyzed (Participants) | 384
  W48 Depression | -1.5 (3.31)
  W72 Depression: number analyzed (Participants) | 214
  W72 Depression | -1.7 (3.19)
Statistical Analysis 1: Comparison: All Patients; Test type: Superiority; p < .0001, Wilcoxon (Mann-Whitney) — All time points

7. Secondary Outcome: Correlation Between the Hospital Anxiety and Depression Scale (HADS) and PASI (FAS)
Description: PASI score, HADS questionnaire correlation using Spearman rank correlation coefficient. It was pre-specified that results would be presented for all patients, not by cohort
Time Frame: Baseline up to approximately 72 weeks
Population: Both arms were combined because there is no clinical rationale to show a difference between the cohorts. Cw6 status does not have any impact on anxiety and depression.
Measure: Number; unit: numbers on scores
Arm/Group | All Patients
Number analyzed (Participants) | 431
numbers on scores
  Baseline | 0.02
  Week 16 | 0.19
  Week 24 | 0.18
  Week 48 | 0.21
  Week 72 | 0.32

8. Secondary Outcome: Changes From Baseline in Body Mass Index (Safety Set)
Description: Change in Body mass index from baseline for patients with a value at baseline and the respective post-baseline visit
Time Frame: Baseline up to approximately 72 weeks
Population: Number of patients varied across visits
Measure: Mean (Standard Deviation); unit: kg/m2
Arm/Group | Cw6-positive AIN457 300 mg | Cw6-negative AIN457 300 mg
Number analyzed (Participants) | 185 | 246
kg/m2
  Week 16: number analyzed (Participants) | 163 | 224
  Week 16 | -0.064 (0.7748) | -0.047 (0.9905)
  Week 24: number analyzed (Participants) | 170 | 231
  Week 24 | 0.086 (1.0213) | -0.071 (1.2260)
  Week 48: number analyzed (Participants) | 103 | 141
  Week 48 | 0.302 (1.3474) | -0.052 (1.4991)
  Week 72: number analyzed (Participants) | 29 | 46
  Week 72 | 0.533 (1.8101) | -0.015 (1.8982)

9. Secondary Outcome: Changes From Baseline in Waist Circumference (Safety Set)
Description: Change in waist circumference from baseline for patients with a value at baseline and the respective post-baseline visit
Time Frame: Baseline up to approximately 72 weeks
Population: Number of patients varied across visits
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Cw6-positive AIN457 300 mg | Cw6-negative AIN457 300 mg
Number analyzed (Participants) | 185 | 246
cm
  Week 16: number analyzed (Participants) | 153 | 210
  Week 16 | -0.86 (3.147) | -0.40 (3.006)
  Week 24: number analyzed (Participants) | 154 | 216
  Week 24 | -0.81 (3.689) | -0.73 (4.119)
  Week 48: number analyzed (Participants) | 95 | 131
  Week 48 | -0.76 (4.596) | -0.72 (5.547)
  Week 72: number analyzed (Participants) | 27 | 43
  Week 72 | -1.81 (4.583) | -0.47 (4.501)

10. Secondary Outcome: Changes From Baseline in Weight (Safety Set)
Description: Change in weight from baseline for patients with a value at baseline and the respective post-baseline visit
Time Frame: Baseline up to approximately 72 weeks
Population: Number of patients varied across visits
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Cw6-positive AIN457 300 mg | Cw6-negative AIN457 300 mg
Number analyzed (Participants) | 185 | 246
kg
  Week 16: number analyzed (Participants) | 163 | 224
  Week 16 | -0.20 (2.242) | -0.13 (2.809)
  Week 24: number analyzed (Participants) | 170 | 231
  Week 24 | 0.24 (3.008) | -0.21 (3.572)
  Week 48: number analyzed (Participants) | 103 | 141
  Week 48 | 0.87 (3.909) | -0.15 (4.329)
  Week 72: number analyzed (Participants) | 29 | 46
  Week 72 | 1.40 (4.678) | -0.05 (5.538)

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) are collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV). All AEs reported in this record are from date of First Patient First Treatment until Last Patient Last Visit) up to approximately 72 weeks
Description: Consistent with EudraCT disclosure specifications, Novartis has reported under the Serious adverse events fields "number of deaths resulting from adverse events" all those deaths, resulting from serious adverse events that are deemed to be causally related to treatment by the investigator.
Groups:
- Cw6-Negative AIN457 300 mg: Cw6-Negative AIN457 300 mg
- Cw6-Positive AIN457 300 mg: Cw6-Positive AIN457 300 mg
Arm/Group | Cw6-Negative AIN457 300 mg | Cw6-Positive AIN457 300 mg
All-Cause Mortality (participants affected / at risk) | 2/246 | 0/185
Serious Adverse Events (participants affected / at risk) | 21/246 | 10/185
Other Adverse Events (participants affected / at risk) | 14/246 | 20/185
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cw6-Negative AIN457 300 mg (N=246) | Cw6-Positive AIN457 300 mg (N=185)
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Hepatic lesion (Hepatobiliary disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 3 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Perirectal abscess (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Vulvovaginal candidiasis (Infections and infestations) | 0 | 1
Alanine aminotransferase increased (Investigations) | 2 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 1
Blood bilirubin increased (Investigations) | 2 | 1
Lipase increased (Investigations) | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Enthesopathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Meniscal degeneration (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Depression (Psychiatric disorders) | 0 | 1
Major depression (Psychiatric disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0
Scrotal inflammation (Reproductive system and breast disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory tract irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cw6-Negative AIN457 300 mg (N=246) | Cw6-Positive AIN457 300 mg (N=185)
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 12
Hypertension (Vascular disorders) | 10 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2016-07-22): https://cdn.clinicaltrials.gov/large-docs/61/NCT02394561/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-20): https://cdn.clinicaltrials.gov/large-docs/61/NCT02394561/SAP_001.pdf